CLINICAL TRIAL: NCT04378244
Title: CORONA: A Phase 1/2 Study Using DeltaRex-G Gene Therapy for Symptomatic COVID-19
Brief Title: CORONA: A Study Using DeltaRex-G Gene Therapy for Symptomatic COVID-19
Acronym: CORONA
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Aveni Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF20-203
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; Cytokine Storm; Acute Respiratory Distress Syndrome
Keywords: cyclin G1; gene therapy; activated T cells
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Respiratory Distress Syndrome | interventions — retrovector encoding mutant anti-cyclin G1

STUDY DESIGN:
Intervention Model Description: Sequential assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DeltaRex-G (Experimental): Escalating doses of DeltaRex-G i.v daily for 7 days as follows:
  Dose Level I: 3-6 patients will receive 1 x 10e11 cfu/dose Dose Level II: 3-6 patients will receive 2 x 10e11 cfu/ dose Dose Level III: 3-6 patients will receive 3 x 10e11 cfu/dose
  Interventions: Drug: DeltaRex-G

INTERVENTIONS:
Drug: DeltaRex-G — This is an open label, dose-seeking phase 1/2 study using escalating doses of DeltaRex-G given intravenously for 7 days in a hospital setting.
  The study will employ the standard "Cohort of Three" design (Storer, 1989). Three patients are treated at each dose level with expansion to six patients per cohort if DLT is observed in one of the three initially-enrolled patients at each dose level. If no DLT occurs in 3 patients, escalation to the next dose level will be permitted. The maximum tolerated dose is defined as the highest safely tolerated dose, where not more than one patient experienced DLT, with the next higher dose level having at least two patients who experienced DLT. No intra-patient dose escalation will take place. Patients who do not complete the 7-day treatment will be replaced.
  Other Names: DeltaRex-G Retroviral Vector Encoding a Cyclin G1 Inhibitor

SUMMARY:
COVID-19 is an infectious disease caused by severe acute respiratory syndrome coronavirus 2. COVID-19 causes life threatening complications known as Cytokine Release Syndrome or Cytokine Storm and Acute Respiratory Distress Syndrome. These complications are the main causes of death in this global pandemic. Over 1000 clinical trials are on-going worldwide to diagnose, treat, and improve the aggressive clinical course of COVID-19. The investigators propose the first, and so far, only gene therapy solution that has the potential to address this urgent unmet medical need.

Rationale

1. There are striking similarities between the damaged lung environment of COVID-19 induced ARDS and the tumor microenvironment (exposed collagen from tissue destruction by invading tumor or by the virus-induced immune response, and presence of activated proliferative cells (cancer cells and tumor associated fibroblasts or activated T cells, macrophages and pulmonary fibroblasts in COVID-19);
2. DeltaRex-G is a disease-seeking retrovector encoding a cytocidal dominant negative human cyclin G1 as genetic payload). When injected intravenously, the DeltaRex-G nanoparticles has a navigational system that targets exposed collagenous proteins (XC proteins) in injured tissues (e.g. inflamed lung, kidney, etc.), thus increasing the effective drug concentration at the sites of injury, in the vicinity of activated/proliferative T cells evoked by COVID-19. Our hypothesis is that DeltaRex-G then enters the rapidly dividing T cells and kills them by arresting the G1cell division cycle, hence, reducing cytokine release and ARDS;
3. Intravenous DeltaRex-G has minimal systemic toxicity due to its navigational system (targeting properties) that limits the biodistribution of DeltaRex-G only to areas of injury where exposed collagenous (XC) proteins are abnormally found; and
4. DeltaRex-G is currently available in FDA approved "Right to Try" or Expanded Access Program for Stage 4 cancers for an intermediate size population. To gain this approval, FDA requires DeltaRex-G to have demonstrated safety and efficacy in early clinical trials.

DETAILED DESCRIPTION:
Background and Proposed Research Importance

Coronavirus disease 2019 is an infectious disease caused by severe acute respiratory syndrome coronavirus 2. COVID-19 causes life threatening complications known as Cytokine Release Syndrome or Cytokine Storm and Acute Respiratory Distress Syndrome. These complications are the main causes of death in this global pandemic. Over 1000 clinical trials are on-going worldwide to diagnose, treat, and improve the aggressive clinical course of COVID-19. The investigators propose the first, and so far, only gene therapy solution that has the potential to address this urgent unmet medical need.

Rationale

1. There are striking similarities between the damaged lung environment of COVID-19 induced ARDS and the tumor microenvironment (exposed collagen from tissue destruction by invading tumor or by the virus-induced immune response, and presence of activated proliferative cells (cancer cells and tumor associated fibroblasts or activated T cells, macrophages and pulmonary fibroblasts in COVID-19);
2. DeltaRex-G is a disease-seeking retrovector encoding a cytocidal dominant negative human cyclin G1 as genetic payload. The DeltaRex-G nanoparticles has a navigational system that targets exposed collagenous proteins in injured tissues, thus increasing the effective drug concentration at the sites of injury, in the vicinity of activated/proliferative T cells evoked by COVID-19. The DeltaRex-G then enters the rapidly dividing T cells and kills them by arresting the G1cell division cycle, hence, reducing cytokine release;
3. Intravenous DeltaRex-G has minimal systemic toxicity due to its disease-seeking properties that limits the biodistribution of DeltaRex-G only to areas of injury where exposed collagenous proteins are abnormally found; and
4. DeltaRex-G is currently available in FDA approved "Right to Try" or Expanded Access Program for Stage 4 cancers for an intermediate size population. To gain this approval, FDA requires DeltaRex-G to have demonstrated safety and efficacy in early clinical trials.

Study Design This is a dose-seeking phase 1/2 study using escalating doses of DeltaRex-G given intravenously for 7 days in a hospital setting, with a randomization schema at the MTD.

The study will include up to three cohorts with increasing DeltaRex-G doses as shown below. The study will employ the standard "Cohort of Three" design (Storer, 1989). Three patients are treated at each dose level with expansion to six patients per cohort if DLT is observed in one of the three initially enrolled patients at each dose level. If no DLT occurs in 3 patients, escalation to the next dose level will be permitted. The maximum tolerated dose is defined as the highest safely tolerated dose, where not more than one patient experienced DLT, with the next higher dose level having at least two patients who experienced DLT. No intra-patient dose escalation will take place.

Patients within the same cohort of 3 will be treated in a staggered manner, i.e., the next subject will receive the product only after the previous subject has completed administration of all doses and has been evaluated on Day 14 (or one week after last DeltaRex-G infusion) to assess safety. At the MTD, after 3 subjects in same cohort have been evaluated with no DLT, subjects in the same cohort may be treated simultaneously.

Patients who do not complete the 7-day treatment will be replaced except if patient developed DLT.

Randomization Schema:

At the highest dose level or when MTD is determined, nine (9) additional patients will be randomized to the treatment arm + standard of care (SOC) vs. standard of care alone (n = 6 patients DeltaRex-G and 3 SOC in each group). Patients will be matched according to symptomatology (e.g. SpO2 >94% at the time of screening), age (within 10 years or at least less than or greater than 65 years), race (black vs non-black), and gender.

Dose of DeltaRex-G: Escalating doses of DeltaRex-G i.v daily for 7 days:

Number of Pts. Dose Level Dose, cfu Max.Volume/24 hrs

3-6 I 1 x 10e11 200 ml 3-6 II 2 x 10e11 200 ml 3-6 III 3 x 10e11 200 ml

Monitoring Plan:

Patient's clinical status including need or duration of mechanical ventilation therapy, change in oxygen saturation, blood counts, lung, liver and kidney function and vital signs, proinflammatory cytokines, including IL-6, IL-12, and tumor necrosis factor α, CRP, LDH, D-Dimer, serum ferritin, chest X-ray are monitored as specified in the protocol and as needed in hospitalized patients during the treatment period, one week later, and every month for 6 months.

Analysis of Primary Endpoint Safety analysis will be performed. The study will employ the standard "cohort of three" design. Three patients are treated at each dose level with expansion to six patients per cohort if DLT is observed in one of the three initially-enrolled patients at each dose level. The maximum tolerated dose is defined as the highest safely tolerated dose, where not more than one patient experienced DLT, with the next higher dose level having at least two patients who experienced DLT. No intra-patient escalation will take place.

Dose limiting toxicity, maximum tolerated dose, incidence and severity of adverse events and significant laboratory abnormalities is the primary endpoint. Safety analysis will be performed on all patients.

Patient incidence of all treatment-related AEs will be tabulated by system organ class and preferred term. Tables of fatal adverse events, serious adverse events, treatment-related AEs, and adverse events leading to withdrawal from investigation product will also be provided. Summary statistics will be provided for total number of doses, average dose administered, and duration of each treatment.

Analysis of Secondary Endpoint Efficacy analysis will be conducted. Change in clinical status such as duration of fever, respiratory destress, pneumonia, cough, sneezing, diarrhea will be documented. ECOG score, mortality, length of hospital stay, duration of respirator therapy, duration of intensive care unit stay, and changes in cytokine pattern will be compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the inclusion criteria in order to be eligible to participate in the study, as follows:

* Male or female ≥ 18 years of age
* Confirmed COVID-19 positive by viral RT PCR
* Patients with severe disease as evidenced by presence of pneumonia, diagnosis of ARDS in hospitalized patients
* Ability to understand the purposes and risks of the study and has signed and dated a written informed consent form approved by the investigator's IRB/Ethics Committee
* Willingness to comply with all study procedures and availability for the duration of the study.
* Adequate hematologic, renal or hepatic function defined by any of the following screening laboratory
* Values:

  i) Neutrophils >1000/uL ii) Platelets > 75,000/uL iii) Serum creatinine <1.5 x ULN or creatinine clearance < 60 mL/min (using the Cockcroft Gault formula) iv) AST/ALT, alk phos <3 x ULN vi) Total Bilirubin <1.5 x ULN
* All women of childbearing potential must have a negative pregnancy test and all subjects must agree to use highly effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 2 months after the last dose.

Exclusion Criteria:

All individuals meeting any of the exclusion criteria at baseline will be excluded from study participation, as follows:

* Females who are pregnant or breast-feeding
* Unwillingness or inability to comply with the study protocol for any reason

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-12 (Estimated); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-07-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 3 weeks
  The study will employ the standard "cohort of three" design (Storer, 1989). Three patients are treated at each dose level with expansion to six patients per cohort if DLT is observed in one of the three initially-enrolled patients at each dose level. The maximum tolerated dose is defined as the highest safely tolerated dose, where not more than one patient experienced DLT, with the next higher dose level having at least two patients who experienced DLT. No intra-patient escalation will take place.

SECONDARY OUTCOMES:
Survival | 2 months
  Duration of survival
Hospital Stay | 3 weeks
  Time of hospital admission to time of discharge
Ventilator Therapy | 3 weeks
  Time from start of mechanical ventilation to extubation or death
Intensive Care Unit Stay | 3 weeks
  Time from start of intensive care to discarge to regular room
Cytokine Pattern | 3 weeks
  Improvement in serum cytokine IL-6, IL12, TNF alpha

CONTACTS AND LOCATIONS:
Overall Officials: Sant P Chawla, MD, Principal Investigator — Mission Community Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behrens A, Gordon EM, Li L, Liu PX, Chen Z, Peng H, La Bree L, Anderson WF, Hall FL, McDonnell PJ. Retroviral gene therapy vectors for prevention of excimer laser-induced corneal haze. Invest Ophthalmol Vis Sci. 2002 Apr;43(4):968-77. PMID 11923236
- [Background] Chawla SP, Chua VS, Fernandez L, Quon D, Saralou A, Blackwelder WC, Hall FL, Gordon EM. Phase I/II and phase II studies of targeted gene delivery in vivo: intravenous Rexin-G for chemotherapy-resistant sarcoma and osteosarcoma. Mol Ther. 2009 Sep;17(9):1651-7. doi: 10.1038/mt.2009.126. Epub 2009 Jun 16. PMID 19532136
- [Background] Gordon EM, Zhu NL, Forney Prescott M, Chen ZH, Anderson WF, Hall FL. Lesion-targeted injectable vectors for vascular restenosis. Hum Gene Ther. 2001 Jul 1;12(10):1277-87. doi: 10.1089/104303401750270931. PMID 11440621
- [Background] Chawla SP, Bruckner H, Morse MA, Assudani N, Hall FL, Gordon EM. A Phase I-II Study Using Rexin-G Tumor-Targeted Retrovector Encoding a Dominant-Negative Cyclin G1 Inhibitor for Advanced Pancreatic Cancer. Mol Ther Oncolytics. 2018 Dec 14;12:56-67. doi: 10.1016/j.omto.2018.12.005. eCollection 2019 Mar 29. PMID 30705966
- [Background] Gordon EM, Hall FL. Rexin-G, a targeted genetic medicine for cancer. Expert Opin Biol Ther. 2010 May;10(5):819-32. doi: 10.1517/14712598.2010.481666. PMID 20384524
- [Background] Hall FL, Gordon EM, Wu L, Zhu NL, Skotzko MJ, Starnes VA, Anderson WF. Targeting retroviral vectors to vascular lesions by genetic engineering of the MoMLV gp70 envelope protein. Hum Gene Ther. 1997 Dec 10;8(18):2183-92. doi: 10.1089/hum.1997.8.18-2183. PMID 9449372
- [Background] Wu L, Liu L, Yee A, Carbonarohall D, Tolo V, Hall F. Molecular-cloning of the human cycg1 gene encoding a g-type cyclin - overexpression in human osteosarcoma cells. Oncol Rep. 1994 Jul;1(4):705-11. doi: 10.3892/or.1.4.705. PMID 21607426
- [Background] Xu F, Prescott MF, Liu PX, Chen ZH, Liau G, Gordon EM, Hall FL. Long term inhibition of neointima formation in balloon-injured rat arteries by intraluminal instillation of a matrix-targeted retroviral vector bearing a cytocidal mutant cyclin G1 construct. Int J Mol Med. 2001 Jul;8(1):19-30. doi: 10.3892/ijmm.8.1.19. PMID 11408944
- [Background] Zhu NL, Wu L, Liu PX, Gordon EM, Anderson WF, Starnes VA, Hall FL. Downregulation of cyclin G1 expression by retrovirus-mediated antisense gene transfer inhibits vascular smooth muscle cell proliferation and neointima formation. Circulation. 1997 Jul 15;96(2):628-35. doi: 10.1161/01.cir.96.2.628. PMID 9244236
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Wu KJ, Yee A, Zhu NL, Gordon EM, Hall FL. Characterization of differential gene expression in monkey arterial neointima following balloon catheter injury. Int J Mol Med. 2000 Oct;6(4):433-40. PMID 10998433
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651